CLINICAL TRIAL: NCT04222608
Title: BRAzilian Registry of Acute Coronary Syndrome in Oncologic Patients - The BRAvAdO Registry
Brief Title: The BRAvAdO Registry
Acronym: BRAvAdO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Instituto do Cancer do Estado de São Paulo (Other); Beneficência Portuguesa de São Paulo (Other); Instituto de Cardiologia do Rio Grande do Sul (Other); InCor Heart Institute (Other)
Responsible Party: Sponsor
Other Study IDs: BRAvAdO
Record Dates: First submitted 2019-11-13; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2019-11

CONDITIONS: ACS - Acute Coronary Syndrome; Oncology
Keywords: Cardio-Oncology; Interventional Cardiology; Cancer; Oncology; Acute Coronary Syndrome; Myocardial Infarction
MeSH Terms: conditions — Acute Coronary Syndrome; Neoplasms; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The BRAVADO Registry pretends to identify stratification, diagnosis, total atherosclerotic burden and treatment approaches in oncologic patients with Acute Coronary Syndrome (ACS) and identify strategies to improve health care quality

ELIGIBILITY:
Inclusion Criteria:

* Definitive cancer diagnosis - biopsy
* Acute Coronary Syndrome - requiring urgent invasive risk stratification

Exclusion Criteria:

* KPS < 60 , ECOG >/ 3
* Life expectancy less 24hs
* End of Life Care
* Lack of consistent record data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with Acute Coronary Syndrome (ACS)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 30 days
  Composite endpoint of All-cause Death, Myocardial Infarction, Stroke and Myocardial Revascularization
Total Atherosclerotic burden and lesion complexity on angiography | 30 days
  The number and location of coronary lesions with obstructions greater than 50% were recorded. Each lesion was classified based on Ambrose's, Goldstein complexity, Leaman and SYNTAX scores.
Incidence of Major Bleeding | 30 days
  Requiring a transfusion of ≥2 U PRBCs Resulting in a decrease in hematocrit of ≥10% Occurring intracerebrally Resulting in stroke or death

CONTACTS AND LOCATIONS:
Locations (1):
- Carlos M Campos, São Paulo, Brazil